CLINICAL TRIAL: NCT06585800
Title: Exploring the Landscape of Somatic Mutations in Human Tissue
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 248671
Record Dates: First submitted 2024-07-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Somatic Mutation
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Collection of blood and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 1.Undergoing surgery: For participants undergoing surgery, research tissue specimens will be sampled from resected tissue - no additional solid tissue research samples will be removed from patients undergoing surgery. Samples taken from surgery will be either from the margins of the resected specimen, or the specimen itself. However this will be done only with agreement with the clinical team and the histopathologist to ensure that clinical pathology is not affected.
  Interventions: Other: sample collection
- 2.1. Undergoing Invasive Procedures (Endoscopy): Endoscopy (oesophagogastroduodenoscopy, small bowel enteroscopy, colonoscopy, sigmoidoscopy, proctoscopy) for suspected gastrointestinal disease e.g. coeliac disease or for surveillance of known conditions/ diseases. For participants undergoing endoscopy as part of their routine clinical care, additional tissue biopsies will be taken for the purpose of this study only in cases where it is safe to do so.
  Interventions: Other: sample collection
- 2.2. Undergoing Invasive Procedures (Biopsy): Tissue Biopsies of solid organs. For participants undergoing tissue biopsy as part of their routine clinical care, additional tissue biopsies will be taken for the purpose of this study only in cases where it is safe to do so. For those undergoing high risk biopsies, e.g. liver biopsies, samples for research will only be taken from clinical specimens, i.e. no additional specimens will be taken solely for the purpose of research.
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — blood and/or tissue collection

SUMMARY:
Every cell in the human body contains a blueprint of the body called the genome. Throughout life, the genome can become damaged resulting in errors (mutations) that can change the way cells behave and may result in diseases such as cancer. Examining the mutations found the genome of both normal (non-cancerous) and diseased cells can give a valuable insight into the very earliest stages of cancer development.

Comparing the number and type of mutations in different normal tissues is revealing new insights, helping us to better understand more about why cancer develops.

DETAILED DESCRIPTION:
The investigators are seeking to characterise somatic mutations found in normal human tissue, as well as diseased tissue. These experiments have shown that a number of mutational processes previously observed in cancer cells, may also be present in normal tissues. By further exploring normal tissue samples from across the body, the investigators will be able to better understand why certain organs are more susceptible to mutations and what underlies the mutational processes active in many different tissue types.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing surgery
* Individuals undergoing invasive procedures, e.g.
* Endoscopy (oesophagogastroduodenoscopy, small bowel enteroscopy, colonoscopy, sigmoidoscopy,proctoscopy) for suspected gastrointestinal disease, e.g. coeliac disease or for surveillance of known conditions/diseases.
* Tissue biopsy - of solid organs
* Prospective sampling will be carried out with the research participants' consent.

Exclusion Criteria:

* where consent has not been received

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Normal (healthy) tissue - across ages 18 - 80+ years
  2. Normal (healthy) tissue, diseased tissue and neoplastic tissue in patients with conditions associated with known disease processes, including syndromes caused by DNA repair defects
  3. Normal (healthy) and neoplastic tissue in patients previously treated with treatments known to cause somatic mutations, e.g. chemotherapy.
  Clinical collaborators will identify and recruit prospective research participants into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of somatic mutation burden | 6.25 years
  Identify and quantify variations that may contribute to disease development and progression between samples from the same donor and different donors, encompassing both healthy individuals and those with diseases.

SECONDARY OUTCOMES:
Number of Somatic Mutations | 6.25 years
  Quantification of the total number of somatic mutations present in the tissue samples.
Spectrum of Mutational Signatures | 6.25 years
  Analysis of the spectrum of mutational signatures, including:
  * Base Substitutions
  * Indels (Insertions and Deletions)
  * Genome Rearrangements
  * Copy Number Changes
Size of Clonal Populations | 6.25 years
  Measurement of the size of clonal populations within the tissue samples.
Relatedness of Clonal Populations | 6.25 years
  Analysis of the genetic relatedness of clonal populations within the tissue samples.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Stratton, Principal Investigator — Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom